CLINICAL TRIAL: NCT02265991
Title: Prospective Biomechanical Analysis of Donor-site Morbidity Following Microvascular Fibula Transplantation in 27 Consecutive Cases: a Clinical Cohort Study.
Brief Title: Prospective Biomechanical Analysis of Donor-site Morbidity Following Microvascular Fibula Transplantation
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Carsten Rendenbach, Resident, Researcher, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: UKEppendorfMKG
Record Dates: First submitted 2014-10-07; First posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Fibula Explantation — surgical harvest of an osteomyocutaenous transplant consisting of a part of the fibula and surrounding soft tissues
  Other Names: Free fibula flap; autologous fibula transfer

SUMMARY:
Pre- and postoperatively patients who underwent free fibula flap were examined regarding donor-site morbidity of the lower extremities.

DETAILED DESCRIPTION:
27 patients are examined before and after microsurgical fibula flap performed at the Department of Oral and Maxillofacial Surgery, University Medical Center Hamburg Eppendorf, Germany.

ELIGIBILITY:
Inclusion Criteria:

* Planned continuity interrupting mandible resection
* Planned mandible reconstruction with free fibula flap
* Informed consent
* Procedure performed at University Medical Center Hamburg Eppendorf

Exclusion Criteria:

* Preexisting pathology/disease of the lower limbs or back (angiologic, neurologic, orthopedic)
* Musculosceletal pain at the time of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with informed consent and that will undergo mandible resection and reconstruction via free fibula flap at the Department of Oral and Maxillofacial Surgery, University Medical Center Hamburg Eppendorf, Germany.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2011-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in Esslinger Fitness Index | 1 day before fibula transplantation and 8.3 months postoperatively on average
  Jumping Mechanography, Functional Assessment on Leonardo Mechanograph GFRP

SECONDARY OUTCOMES:
AOFAS Score | 1 day before fibula transplantation and 8.3 months postoperatively on average
  Objective and Subjective Score for functionality and pathology of the ankle region
Balance Test | 1 day before fibula transplantation and 8.3 months postoperatively on average
  Functional Assessment on Leonardo Mechanograph GFRP, measures the patients' stability
Range of Motion | 1 day before fibula transplantation and 8.3 months postoperatively on average
  Measuring Ankle Motion before and after surgery with a goniometer